CLINICAL TRIAL: NCT00719641
Title: A Trial of Segmental Stiffening Wires to Improve the Efficiency and Patient Tolerability of Colonoscopy
Brief Title: Experimental Device to Improve Colonoscopy
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080173; 08-DK-0173
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2019-10

CONDITIONS: Colonoscopy; Looping; Prevent Looping; Colon Cancer Screening
Keywords: Colonoscopy; Looping; Prevent Looping; Colon Cancer Screening; Segmental Stiffening Wire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (4):
- Phase 1: Single Colonoscopy: Feasibility testing using the segmental stiffening wire
- Phase 2; Not randomized: Phase 2 participants who did not have looping during first colonoscopy
- Phase 2: Randomized to SSW during first colonoscopy: Phase 2 participants in whom looping occurred on first biopsy, randomized to subsequent use of segmental stiffening wire, then colonoscopy with no segmental stiffening wire upon repeat colonoscopy the next day.
- Phase 2: Randomized to SSW during second colonoscopy: Phase 2 participants in whom looping occurred on first biopsy, randomized to no subsequent use of the segmental stiffening wire that day, then colonoscopy with segmental stiffening wire upon repeat colonoscopy the next day.

SUMMARY:
This study will test the use of a new device called a segmental stiffening wire (SSW) in colonoscopy to correct a problem called looping. Colonoscopy is the best test for detecting early colon cancer and removing growths called polyps, which can become colon cancer. Sometimes the flexible tube (colonoscope) used in the procedure loops at a certain point as it advances through the colon, making it difficult to move further and causing the patient pain from excessive stretching of the colon. The SSW is designed to prevent this by stiffening the part of the tube that would otherwise form the loop.

Healthy subjects between 50 and 80 years of age and healthy subjects 40 years and older who have a family history of colon cancer may be eligible for this study.

Participants undergo colonoscopy a day after self-administering a bowel cleansing preparation. The first part of the procedure is done similarly to that of a flexible sigmoidoscopy, and no sedation or pain medication is used. The colonoscope is inserted into the rectum and advanced about one-third the length of the colon. Pain or discomfort should be mild to moderate cramping and a feeling of having to move the bowels. The subject is asked to score his or her pain level at this point using a standard pain scale. If there is pain, the procedure is stopped and an x-ray is taken to determine if the colonoscope has looped. If it has, the loop is undone and the SSW is used. Another x-ray is then taken to document that the loop has been prevented with the SSW, and the procedure is completed as per standard medical practice. Subjects are taken to the recovery area, informed of the test results and then discharged home in the care of an accompanying adult.

DETAILED DESCRIPTION:
Colonoscopy can be challenging to perform and painful due to looping of the colonoscope. Looping occurs when further insertion of the colonoscope results in a loop forming in the shaft of the colonoscope instead of advancement of the tip. Attempts have been made to solve this problem, but to date there is no perfect solution. Since colonoscopy is the gold standard for colon cancer screening providing a device that could prevent looping would be valuable. We have developed an experimental device that has not been approved outside of the context of this study known as the Segmental Stiffening Wire (SSW). This wire will be utilized by passing it through the biopsy channel of the endoscope. The wire has a 15-25 inch area of increased thickness and stiffness. The stiffened section can be advanced into areas of looping in an effort to prevent re-looping. We will conduct a pilot study in two phases. The first phase will include approximately 10 healthy volunteers who will undergo colonoscopy using the SSW. Fluoroscopy will be used to determine if the device prevents re-looping. If in phase 1 the device is successful in over 30% of episodes, the second phase will be undertaken. In the second phase volunteers willing to undergo two colonoscopies on consecutive days will be recruited. Volunteers who experience looping will be randomized as to whether the SSW is available. These volunteers will then undergo an otherwise identical colonoscopy on the following day except the SSW will be available if it was not on the first colonoscopy or it will not be available if it was on the first colonoscopy. Volunteers who undergo two colonoscopies will not need a second bowel preparation but will be maintained on a clear liquid diet between the two procedures. Volunteers in which looping does not occur will have their initial colonoscopy completed as normal and then will leave the study. If unable to obtain sufficient volunteers willing to undergo dual colonoscopy, then volunteers willing to undergo single colonoscopy will be included and their procedures will be done with or without the SSW in random fashion. The endpoints will be cecal intubation time; cecal intubation rate; quantity of sedation/analgesia; number of ancillary maneuvers; pain/sedation as measured by the Visual Analog Pain Scale, the Ramsey Sedation Scale, and clinical observations; vital sign changes; and the endoscopists subjective assessment of procedure difficulty and the usefulness of the SSW.

ELIGIBILITY:
* INCLUSION CRITERIA:

Colonoscopy is indicated based on well-established national guidelines. This includes volunteers age 50 or greater who are at average risk for colon cancer, and volunteers age 40 or greater who are at increased risk based on a personal history of colon polyps or a family history of colon polyps or cancer.

Volunteer meets the criteria of Anesthesia Level 1 or 2.

Volunteer agrees to undergo the study procedures.

EXCLUSION CRITERIA:

Ongoing psychiatric history including volunteers who have been hospitalized for psychiatric reasons, have missed significant number of days of work for psychiatric reasons, or who admit to suicidal ideations.

Former or current history of alcohol or drug dependency.

History of colonic resection.

Pregnancy.

Age greater than 80 or less than 40.

Prior radiation to the abdomen or pelvis.

American Society of Anesthesiologists Grade 3, 4, or 5.

Allergy or other contraindications to midazolam or fentanyl.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects between 50 and 80 years of age and healthy subjects 40 years and older who have a family history of colon cancer may be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-08-05 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
Cecal Intubation Time | During colonoscopy, up to 60 minutes
  Cecal intubation time of colonoscopy with SSW, compared to without SSW
Number of Participants Without Re-looping Among Those With Looping | During the colonoscopy, up to 60 minutes
  Re-looping during the procedure that used SSW, this information only collected when using SSW

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Wank, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Meissner HI, Breen N, Klabunde CN, Vernon SW. Patterns of colorectal cancer screening uptake among men and women in the United States. Cancer Epidemiol Biomarkers Prev. 2006 Feb;15(2):389-94. doi: 10.1158/1055-9965.EPI-05-0678. PMID 16492934
- [Background] Kahi CJ, Rex DK. Current and future trends in colorectal cancer screening. Cancer Metastasis Rev. 2004 Jan-Jun;23(1-2):137-44. doi: 10.1023/a:1025871231346. PMID 15000154
- [Background] Wu GH, Wang YM, Yen AM, Wong JM, Lai HC, Warwick J, Chen TH. Cost-effectiveness analysis of colorectal cancer screening with stool DNA testing in intermediate-incidence countries. BMC Cancer. 2006 May 24;6:136. doi: 10.1186/1471-2407-6-136. PMID 16723013
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-DK-0173.html